CLINICAL TRIAL: NCT05709509
Title: Effect of Colchicine in Regulating MMP-9, NOX-2, and TGF- β1 After Myocardial Infraction in Stable Patients
Brief Title: Effect of Colchicine on MMP-9, NOX2, and TGF-β1 in Myocardial Infarct
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RSD dr. Soebandi (Other Government)
Collaborators: Universitas Jember (Unknown); University of Brawijaya (Other)
Responsible Party: Principal Investigator, Suryono Suryono, Principal Investigator, RSD dr. Soebandi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: colchicine and Cardiovascular
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: ST Elevation Myocardial Infarction; Colchicine; Cardiac Remodeling, Ventricular
Keywords: STEMI; Colchicine; MMP-9; NOX2; TGF-beta 1
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Ventricular Remodeling; Camurati-Engelmann Syndrome | interventions — Colchicine; Percutaneous Coronary Intervention; Aspirin; Nitrates

STUDY DESIGN:
Intervention Model Description: All subjects were allocated to 4 different groups: Late PCI + Colchicine, Late PCI + Optimal Medical Treatment, Optimal Medical Treatment + Colchicine, and Optimal Medical Treatment Only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Late PCI + Colchicine (Experimental): Subjects that undergo late PCI (12-48 hours after STEMI), received optimal medical treatment (statin, aspirin, P2Y12 inhibitor, and nitrate), and colchicine
  Interventions: Drug: Colchicine; Procedure: Percutaneous Coronary Intervention; Other: Optimal medical treatment including statin, aspirin, P2Y12 inhibitor, and nitrate.
- Late PCI + Optimal Medical Treatment (Experimental): Subjects that undergo late PCI (12-48 hours after STEMI) and received optimal medical treatment (statin, aspirin, P2Y12 inhibitor, and nitrate)
  Interventions: Procedure: Percutaneous Coronary Intervention; Other: Optimal medical treatment including statin, aspirin, P2Y12 inhibitor, and nitrate.
- Optimal Medical Treatment + Colchicine (Experimental): Subjects that received optimal medical treatment (statin, aspirin, P2Y12 inhibitor, and nitrate) and colchicine
  Interventions: Drug: Colchicine; Other: Optimal medical treatment including statin, aspirin, P2Y12 inhibitor, and nitrate.
- Optimal Medical Treatment (Placebo Comparator): Subjects that received optimal medical treatment (statin, aspirin, P2Y12 inhibitor, and nitrate)
  Interventions: Other: Optimal medical treatment including statin, aspirin, P2Y12 inhibitor, and nitrate.

INTERVENTIONS:
Drug: Colchicine — Colchicine: A major alkaloid from Colchicum autumnale L. and found also in other Colchicum species. commonly used as anti-inflammatory drugs.
  Arms: Late PCI + Colchicine; Optimal Medical Treatment + Colchicine
Procedure: Percutaneous Coronary Intervention — Percutaneous Coronary Intervention: a family of minimally invasive procedures used to open clogged coronary arteries (those that deliver blood to the heart)
  Arms: Late PCI + Colchicine; Late PCI + Optimal Medical Treatment
Other: Optimal medical treatment including statin, aspirin, P2Y12 inhibitor, and nitrate. — The subjects just received optimal medical treatment including statin, aspirin, P2Y12 inhibitor, and nitrate.
  Other Names: No Intervention

SUMMARY:
Reducing NOX-2, MMP-9, and TGF-β1 Expression in Preventing Ventricular Remodelling Post Acute ST-Segment Elevation Myocardial Infarction using Colchicine (Post Late Reperfusion Percutaneous Coronary Intervention and Non-Reperfusion and In Vitro Study on Ischemic Rat Cardiomyocyte Culture Model). Coronary heart disease (CHD) is the most common cause of mortality and disability worldwide. The handling of reperfusion in Indonesia is still far below the required standard. Most STEMI patients in Indonesia arrive late to a health facility with symptoms that have been present for more than 12 hours (late-onset). Heart failure following a myocardial infarction is one of the long-term complications of STEMI. Patients with STEMU who do not receive reperfusion were more likely to develop this consequence. According to several studies, microtubules in cardiomyocytes have been identified as an essential regulator of cardiomyocytes' ability to respond to shear stress, which offers compression resistance and facilitates mitochondrial energy production. Microtubule densification, which occurs due to remodelling in heart failure, disrupts the microtubule network. The role of reactive oxygen species (ROS) produced by ischemic myocardium in this remodelling is thus inextricably linked. NADPH oxidase is one of the enzymes involved (NOX). NOX-2 levels have been reported to be higher in myocardial infarction and cardiac remodelling, and it has a close interaction with microtubule network, with damage of microtubule tissue increasing NOX-2 generation of reactive oxygen species. By eroding the ECM and triggering cytokines and chemokines to recruit inflammatory cells to eliminate necrotic cardiomyocytes, matrix metalloproteinase 9 (MMP-9) aids tissue rebuilding. Induction and activation of endogenous TGF-signaling pathways after myocardial infarction have also been discovered to play a function. TGF-β may play a role in the resolution of the inflammatory response in the early stages of infarct repair by inactivating macrophages and decreasing endothelial cell chemokine and cytokine production. TGF-β stimulates the fibrogenic pathway by causing extracellular matrix deposition and fibrosis later. Colchicine is a commonly prescribed anti-inflammatory medication with a low cost. the mechanism of colchicine is tubulin binding, which prevents microtubule assembly and polymerization. Colchicine inhibits microtubule development at low concentrations and promotes microtubule depolymerization at higher concentrations. Several studies have demonstrated that low-dose colchicine can help reduce severe cardiac outcomes such as cardiovascular mortality, stroke, and cardiac arrest following myocardial infarction. Colchicine is known to cause partial restoration of microtubule tissue in the perinuclear region. Colchicine has also been shown in earlier research to reduce the expression of MMP-9, NOX2, and TGF-β This study aims to evaluate whether colchicine could prevent ventricular remodelling in STEMI patients with delayed reperfusion and non reperfusion. The minor hypothesis of this study was colchicine can lower NOX-2, MMP-9, and TGF-β expression in the clinical situation of patients with delayed and non-reperfusion STEMI following PCI. Randomization with 1:1 allocation were used to classify the patients, each group include 41 patients with one group receiving colchicine therapy and standard therapy and the other receiving standard therapy only. Colchicine administration was the independent variable. STEMI patients with delayed and non-reperfusion IKP who met the inclusion criteria are included in this randomized clinical trial. Left ventricular end-diastolic volume (LVEDV) was the dependent variable while serum MMP-9, NOX-2, and TGF-β were the intermediate variables. In the treatment group, colchicine 1 mg is administered before PCI or admission to the ICCU, and colchicine is continued at 0.5 mg/day for a month. Within 24 to 36 hours of treatment initiation, the patient had echocardiography, NOX-2, MMP-9, and TGF-β levels evaluated. On days 4-5, a second NOX-2, MMP-9, and TGF-β screening were performed. The follow up two months after treatment initiation includes an assessment of drug compliance, symptoms, and echocardiography. Depending on the normality of the data distribution, the difference between groups is performed using the unpaired T-test or the Mann-Whitney test. The significant difference between the treatment groups is indicated by a p-value of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who presenting with STEMI more than 12 hours from the onset of chest pain
* Aged 40-70 years
* Agreed with the informed consent

Exclusion Criteria:

* aged <40 or >70 years
* subjects that have unstable condition such as comorbid disease (infection, inflammation, malignancy, severe renal failure (EGFR <30), a history of hepatic cirrhosis, acute exacerbation of hepatitis, or severe liver disease, alcoholic patient, cardiac arrest, ventricular fibrillation or cardiogenic shock, unstable hemodynamic)
* subjects that have colchicine hypersensitivity
* pregnancy or breastfeed

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
The change between 24 hours MMP-9 to day 5 | 24 Hours, Day 5
  Matrix metallopeptidase 9 (MMP-9), also known as 92 kDa type IV collagenase, 92 kDa gelatinase or gelatinase B (GELB), is a matrixin, a class of enzymes that belong to the zinc-metalloproteinases family involved in the degradation of the extracellular matrix.
The change between 24 hours NOX2 to day 5 | 24 Hours, Day 5
  NADPH oxidase 2 (Nox2), also known as cytochrome b(558) subunit beta or Cytochrome b-245 heavy chain, is a protein that in humans is encoded by the NOX2 gene (also called CYBB gene). The protein is a superoxide generating enzyme which forms reactive oxygen species (ROS).
The change between 24 hours TGF-β1 to day 5 | 24 Hours, Day 5
  Transforming growth factor β1 (TGFB1) is a multifunctional secreted protein that generally regulates immune function,544 as well as cell survival and migration, through the Sma- and Mad-related proteins (SMAD) signaling pathway.
Left ventricular end-diastolic volume (LVEDV) | Month 1
  The volume of blood in the left ventricle at the end of ventricular filling is called the end-diastolic volume (EDV), which is about 120 mL in the adult human.

SECONDARY OUTCOMES:
Number of subjects with hypertension | Baseline
  Hypertension is defined as a systolic blood pressure (SBP) of 140 mm Hg or more, or a diastolic blood pressure (DBP) of 90 mm Hg or more
Number of subjects with diabetes | Baseline
  History of diabetes is defined as having fasting blood glucose 126 mg/dL or HBA1c >6.5%
Smoking status among the subjects | Baseline
  Smoking or Ex-smoking
Number of subjects with dyslipidemia | Baseline
  Dyslipidemia is the imbalance of lipids such as cholesterol, low-density lipoprotein cholesterol, (LDL-C), triglycerides, and high-density lipoprotein (HDL)
Type of infark among the subjects | Baseline
  Type of infark (large or small) that happen to the subjects

CONTACTS AND LOCATIONS:
Locations (1):
- RSD dr Soebandi, Jember, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided